CLINICAL TRIAL: NCT05922137
Title: Oriental Intervention for Enhanced Neurocognitive Health (ORIENT) Diet in Patients With Intracranial / Carotid Stenosis : a Randomized Controlled Trial
Brief Title: Oriental Intervention for Enhanced Neurocognitive Health (ORIENT) Diet in Patients With Intracranial / Carotid Stenosis
Acronym: ORIENT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ORIENT-ICS
Record Dates: First submitted 2023-05-07; First posted 2023-06-28 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2024-09

CONDITIONS: Cognitive Decline; Cognitive Change; Stenosis; Dementia
Keywords: Cognitive decline
MeSH Terms: conditions — Cognitive Dysfunction; Constriction, Pathologic; Dementia | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Diet advice (Placebo Comparator): Usual diet advice + standard medical treatment
  Interventions: Behavioral: Usual Diet advice
- ORIENT diet intervention (Active Comparator): 6 month intervention of ORIENT diet + standard medical treatment
  Interventions: Behavioral: Oriental Intervention for Enhanced Neurocognitive Health (ORIENT) diet

INTERVENTIONS:
Behavioral: Usual Diet advice — The usual diet advice include recommendations in guidelines, such as reducing salt and limiting alcohol consumption
  Arms: Usual Diet advice
Behavioral: Oriental Intervention for Enhanced Neurocognitive Health (ORIENT) diet — The ORIENT diet has the same basic components of the Dietary Approaches to Stop Hypertension (DASH), Mediterranean and MIND diets, but uniquely adjusting some of components according to the evidence derived from Asian prospective cohorts and the Chinese eating habits.
  Arms: ORIENT diet intervention

SUMMARY:
To test the effects of 6 month additional intervention of ORIENT diet versus usual medical treatment for Intracranial / Carotid Stenosis on cognitive decline, multi-mode MRI image markers and serum and fecal biomarkers in a randomized controlled trial of 120 patients with intracranial / carotid stenosis, who are aged older than 40 years and without dementia.

DETAILED DESCRIPTION:
Oriental Intervention for Enhanced Neurocognitive Health (ORIENT) diet in Patients With Intracranial / Carotid Stenosis is designed to test the impact of a 6-month intervention utilizing a culturally adapted version of the MIND diet, named as the ORIENT diet, on 120 older patients (aged 40 years and above and without dementia) diagnosed with intracranial/carotid stenosis (defined as ≥ 50% stenosis in unilateral intracranial/carotid artery as detected by vascular imaging diagnostic techniques, such as magnetic resonance angiography). The ORIENT diet retains the core components of the DASH, Mediterranean, and MIND diets, but incorporates adjustments according to evidence derived from Asian prospective cohorts and Chinese dietary practices. Participants in the intervention group will receive standard medical treatment in conjunction with the ORIENT diet intervention, while those in the control group will undergo standard medical treatment and receive usual dietary advice. The study's primary objective is to assess the influence of the ORIENT diet on cognitive function and brain macro- and microstructural integrity in patients with intracranial/carotid stenosis. This will be achieved through the administration of neuropsychological assessments and multi-modal magnetic resonance imaging at 6-month intervals until the completion of the trial. The investigation will explore potential mediators and modifiers of the intervention's effects by examining various cardiovascular risk factors, serum and fecal biomarkers, and underlying biological mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 40 years
* ≥ 50% stenosis in unilateral intracranial / carotid artery
* Written informed consent available
* Willingness to complete all assessments and participate in follow-up
* Adequate Visual and auditory acuity to undergo neuropsychological testing

Exclusion Criteria:

* Previous history of major head trauma and any intracranial surgery
* Intracranial abnormalities, such as intracerebral hemorrhage, subarachnoid hemorrhage and other space occupying lesions
* Extrapyramidal symptoms or mental illness which may affect neuropsychological measurement
* Severe loss of vision, hearing, or communicative ability
* Nuts, berries, olive oil, or fish allergies
* Patients presenting a malignant disease with life expectancy < 3 years
* Participation in an ongoing investigational drug study

Exit Criteria:

* Not meet the inclusion criteria
* For any poor adherence, not comply with the requirements of the follow-up, or safety reasons determined by investigator
* Any adverse or serious adverse events during the study period judged by Investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-05-21 (Actual); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Global cognitive function change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol | 6 months
  Primary Outcome

SECONDARY OUTCOMES:
Cognitive domain change assessed with NINDS-CSN protocol, including working memory, executive function, language, visual motor speed, visual spatial function, memory and recognition | 6 months
  short-term secondary outcome
Cognitive function change assessed by Montreal Cognitive Assessment (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 6 months
  short-term secondary outcome
Changes in functional network-related characteristics assessed by functional magnetic resonance imaging (fMRI), including intra- and inter-network connectivity, graph theory, and dynamic functional connectivity | 6 months
  short-term secondary outcome
Changes in white matter hyperintensity (WMH) assessed on MRI with T2-Fluid-Attenuated-Inversion-Recovery (FLAIR) sequence | 6 months
  short-term secondary outcome
Changes in cerebral glymphatic function assessed by non-invasive diffusion tensor image analysis along the perivascular space (ALPS-index) | 6 months
  short-term secondary outcome
Changes in cerebral blood flow (CBF) in the territory of the culprit artery assessed by arterial spin labeling (ASL) perfusion image | 6 months
  short-term secondary outcome
Metabolite composition to measure the metabolite profiles in participants' faecal samples and serum samples | 6 months
  short-term secondary outcome: metabolite composition was analyzed via liquid chromatography tandem mass spectrometry (LC-MS/MS)
Metabolite composition to measure the metabolite profiles in participants' faecal samples and serum samples | 2 years
  long-term secondary outcome: metabolite composition was analyzed via liquid chromatography tandem mass spectrometry (LC-MS/MS)
Gut microbiota determined by measuring specific bacterial levels in the fecal samples | 6 months
  short-term secondary outcome
Gut microbiota determined by measuring specific bacterial levels in the fecal samples | 2 years
  long-term secondary outcome
Incidence of stroke event including ischemic and hemorrhagic stroke | 6 months and 2 years
Change in the Oriental Intervention for Enhanced Neurocognitive Health (ORIENT) diet scale (minimum value = 0, maximum value = 14, and higher scores mean a better outcome) | 6 months
  short-term secondary outcome
Change in the Mediterranean-DASH Diet Intervention for Neurodegenerative Delay (MIND) diet scale (minimum value = 0, maximum value = 15, and higher scores mean a better outcome). | 6 months
  short-term secondary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affilated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China